CLINICAL TRIAL: NCT03493438
Title: The Effect of Different Physiotherapy Interventions on Patients With Chronic Low Back Pain
Brief Title: Different Physiotherapy Interventions on Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, aydan aytar, ASSOC. PROF., Baskent University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA 18/27
Record Dates: First submitted 2018-04-04; First posted 2018-04-10 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Exercise Training
MeSH Terms: interventions — Exercise; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized controled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Relaxation Group (Experimental): Patients performed Jacobson relaxation technique in supine position. Respiration control and various visual imaging techniques were used during the technique. Relaxation exercises were made within the supervision of a physiotherapist. The application period was 20 minutes for one session, 3 days a week and totally six weeks.
  Interventions: Other: exercise
- Proprioceptive Neuromuscular Facilitation Group (Experimental): Patients exercised with proprioceptive neuromuscular facilitation technique for trunk muscles using chopping and lifting patterns with ritmic initiation PNF exercises were made by the physiotherapist. The application period was 20 minutes for one session, 3 days a week and totally six weeks.
  Interventions: Other: exercise
- Core stabilization group (Experimental): Patients had core stabilization exercises that involved spinal mobility. The patients performed the drawing-in maneuver within various visual imaging techniques during all exercises, especially with respiratory control. Exercises were made within the supervision of a physiotherapist. The application period was 20 minutes for one session, 3 days a week and totally six weeks.
  Interventions: Other: exercise
- control group (Other): Patients in the control group were told the importance of a single session exercise
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — A hot pack and conventional transcutaneous electrical stimulation (TENS) will be applied with a Chattanoga Intelect® stimulator for 20 minutes at a frequency of 100 Hz and a transition time of 60 μs. The duration of application was 3 days per week and six weeks for each of the four groups. These practices were also applied to individuals in all four groups.
  Other Names: A hot pack, conventional transcutaneous electrical stimulation (TENS) and exersice

SUMMARY:
Low back pain is an extremely common health problem that most people suffers at any point in their life. Low back pain is the leading cause of activity limitation and work absence throughout much of the world and it causes some economic problems for just not only individuals but also governments. ) The purpose of the study was to investigate the effects of different physical therapy techniques on pain, function and core stability in patients with low back pain.

DETAILED DESCRIPTION:
Low back pain is an extremely common health problem that most people suffers at any point in their life. Low back pain is the leading cause of activity limitation and work absence throughout much of the world and it causes some economic problems for just not only individuals but also governments. Low back pain is a symptom rather than a disease. Non-specific low back pain term is used when the pathoanatomical cause of the pain cannot be determined. Most patients had pain that caused interference with daily function. Low back pain can be triggered by physical factors (eg, lifting awkwardly) or psychosocial factors (eg, being fatigued or tired), or by a combination of the two (eg, being distracted while lifting). There are several nonpharmacologic treatment options that include analgesics, muscle relaxants, physical therapy modalities, spinal manipulative therapy, psychological therapies and others for back pain. Unfortunately, none of the therapies has been established as superior to others. Controversly some of the investigators suggest individuals with chronic LBP can more benefit from exercise therapy interventions but still evidence on the effectiveness of nonpharmacologic therapies was very limited. The purpose of the study was to investigate the effects of different physical therapy techniques on pain, function and core stability in patients with low back pain.

Female patients with chronic, nonspecific LBP who were either undergoing or initiating physical therapy treatment at the Baskent University Ankara Hospital Physical Therapy and Rehabilitation outpatient clinic participated in the study.

Before the study began patients were randomized into four groups: Relaxation, Proprioceptive Neuromuscular Facilitation (PNF), core stability and control groups.

Descriptive characteristic of patients was evaluated at the beginning of the study. Pain, functionality, kinesiophobia and core stability was evaluated before and after the treatments. Pain and functionality were the primer outcome measures of this study, kinesiophobia, core stability and satisfaction were seconder. Patient satisfaction was assessed after the treatments.

A hot pack and conventional transcutaneous electrical stimulation (TENS) will be applied with a Chattanoga Intelect® stimulator for 20 minutes at a frequency of 100 Hz and a transition time of 60 μs. The duration of application was 3 days per week and six weeks for each of the four groups. These practices were also applied to individuals in all four groups.

The program was involved one of the following techniques of relaxation: proprioceptive neuromuscular facilitation: core stability or control. At the end of the treatments, the individuals in each group were given exercise as home brochure.

ELIGIBILITY:
Inclusion Criteria:

* inclusion criteria;

  1. Patients had to have LBP for at least 3 months,
  2. Patients who reported osteoarthritis or disk lesions (without neurologic compromise) with or without leg pain,
  3. Patients between 18 and 65 years of age,

Exclusion Criteria:

* Patients were excluded if they demonstrated any of the following;

  1. They had neurologic signs, specific spinal pathology (eg, malignancy, inflammatory joint disease, bone disease),
  2. They had undergone back and lower extremity surgery.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-06-26 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 6 weeks
  Pain intensity was measured with visual analog scale (VAS). For VAS, it is desirable that patients express their pain with a (X) mark on a scale of 100 mm. According to this, "0" means that the patients have no pain and "100" means that they have worst pain. The distance between the marking point and the start of the line is measured in millimeters and the numerical value found determines the pain intensity of patients. The total pain intensity is measured with the scale of Likert type of 6 points. In this scale "0" indicates no pain and "5" indicates worst pain.
Functionality | 6 weeks
  The Oswestry Low Back Pain Questionnaire was used to assess the functioning of daily living activities in low back pain. There are 10 questions in the questionnaire, 6 options in each question, ranging from 0 to 5 points. The patient is asked to choose the expression that best describes the situation. The highest score was 50, with mild functional impairment between 1-10 points, moderate functional impairment between 11-30 points, and severe functional impairment between 31-50 points. The Turkish version of the questionnaire was validated and reliable.
Kinesiophobia | 6 weeks
  Individuals' kinesiophobia were assessed by using the Tampa Kinesiophobia Scale. The questionnaire is a 17-item measure designed to measure fear of movement / re-injury. The scale includes injury / re-injury and fear-avoidance parameters in work-related activities. A 4-point Likert Scale (1 = strongly disagree, 4 = fully agree) is used on the scale. A total score is calculated after the reversal of 4, 8, 12, and 16 questions. The patient has a total score between 17-68. The high score on the scale indicates that the kinesophobia is also high. The Turkish version of the questionnaire was validated and reliable
core stability | 6 weeks
  Core stability was assessed with the pressure device (Stabilizer Pressure Biofeedback, USA, Chattanooga Group, Hixson, TN). For transversus abdominus (TrA) and multifidus (MF) muscle strength the patients performed the drawing-in maneuver in a supine position, with their knees flexed at 90°. To perform abdominal drawing-in maneuver, all the subjects were instructed to slowly draw in their lower abdomen as if they were holding their urine and then draw up their pelvic floor muscle so that it could contract, together with their lower abdomen, while continuing normal breathing. The end part of the pressure device was placed on the posterior superior iliac spine. The pressure gauge was set to indicate 40 mmHg before the drawing-in maneuver began. The subjects were told to increase the pressure by 10 mmHg using the drawing-in maneuver on the verbal instruction, "start", and to maintain the state for 5 seconds. Pressure changes were recorded as mmHg.

SECONDARY OUTCOMES:
patient satisfaction | 6 weeks
  Patient satisfaction was measured with VAS for pain and functionality. The patients asked to express their satisfaction with a (X) mark on a scale of 10 cm. According to this, "0" means that the patients have worst satisfaction and "100" means that they greatest satisfaction. The distance between the marking point and the start of the line is measured and numerical value taken as a satisfaction level of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided